CLINICAL TRIAL: NCT02847351
Title: A Mild Supplementation of Arabinoxylan Fiber Improves Homa Index in Overweight and Obese Subjects. Results From a Randomized Cross Over Trial.
Brief Title: A Mild Supplementation of Arabinoxylan Fiber Improves Homa Index in Overweight and Obese Subjects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Chiara Muggia; MD, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 30200/9334
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: arabinoxylan, HOMA index, glycemic control, obesity.
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Diet (CD) (Placebo Comparator): Period 1(the first 4 weeks): 10 subjects were randomly assigned to Control Diet: they replaced for 4 weeks all the carbohydrates consumed in day (bread, pasta, runks) with crackers produced with a normal white grain flour. After this period they crossed to period 2 (the second 4 weeks of treatment) without any wash out: they replaced for 4 weeks all the carbohydrates consumed in day (bread, pasta, runks) with crackers produced with Arabinoxylan-enriched flour.
  Interventions: Dietary Supplement: Arabinoxylan Diet
- Arabinoxylan Diet (AXD) (Experimental): Period 1(the first 4 weeks): 9 subjects were randomly assigned to Arabinoxylan-Diet: they replaced for 4 weeks all the carbohydrates consumed in day with crackers baked with an Arabinoxylan-enriched flour. After this period they crossed to period 2 (the second 4 weeks of treatment) without any wash out: they replaced for 4 weeks all the carbohydrates consumed in day with crackers produced with a normal white grain flour
  Interventions: Dietary Supplement: Arabinoxylan Diet

INTERVENTIONS:
Dietary Supplement: Arabinoxylan Diet — 19 free-living subjects (16 F/ 3M) attending from one year the Outpatient Obesity Clinic Policlinico S. Matteo were enrolled. All subjects were already reached weight loss and were in a sort of "weight steady state". Based on 7-day food diary, a nutritionist composed 19 isocaloric diets, replacing all consumed carbohydrates with normal or AX crackers. The mean carbohydrates intake was 189.5g, with total fiber 20.6g. In AX diet total fiber was 25.3g/day (20.6 plus 4.68g of AX).
  Height, weight, waist circumference were obtained at time 0, at week 4 and 8. At every time were collected blood samples for glucose, insulin, total cholesterol, HDL-chol., tryglicerides, plasma acyl and des-acyl ghrelin. Glucose and insulin were , also collected 2 h after a 75 g oral glucose tolerance test (OGTT).
  Other Names: Integralbianco® flour- Farine Varvello

SUMMARY:
The study aimed to investigate whether an Arabinoxylan-enriched crackers consumption for 4 weeks in overweight and obese patients without diabetes mellitus have specific healthy effects on glycemic control (reduction of homeostatic model assessment -HOMA index-). Furthermore, study evaluated the effects of Arabinoxylan on insulin, lipid and Ghrelin.

DETAILED DESCRIPTION:
The beneficial effects of soluble dietary fiber to health are well known: many studies show clearly that it delays the onset of cardiovascular disease and some cancers, and improves glycemic control in type 2 diabetes. (1,2). Overweight and obesity are known to be associated with increased rate of diabetes, hypertension and cardiovascular diseases, as well as to colon and breast cancer. The introduction of 25-30gr of dietary fiber daily would therefore indicated not only in type 2 diabetic subjects, but also in obese and overweight patients. Most of the foods commonly consumed in Western countries are low in dietary fiber: to reach the recommended levels people should introduce whole grain cereals, legumes, vegetables and dried fruits, not always accepted. We tested the effects on health of crackers baked with a special Integralbianco® flour, enriched with 3,2g of Arabinoxylan / 100g (vs refined flour).

ELIGIBILITY:
Inclusion Criteria:

* males and females
* age ≥ 18 years
* Body mass Index ≥ 27

Exclusion Criteria:

* diabetes mellitus
* already established organ damage
* debilitating diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of Homa Index after Ax Diet vs CD Diet | 4 weeks of arabinoxylan dietetic supplementation
  The study aimed to investigate whether an Arabinoxylan enriched crackers consumption for 4 weeks in overweight or obese patients without diabetes mellitus have specific healthy effects on glycemic control, evaluated as reduction of Homa Index.

SECONDARY OUTCOMES:
Improvement of lipidic profile after AxDiet vs CD Diet | 4 weeks of arabinoxylan dietetic supplementation
  The study aimed to investigate whether an Arabinoxylan enriched crackers consumption for 4 weeks had some benefic effects on lipids.
Improvement of weight after AxDiet vs CD Diet | 4 weeks of arabinoxylan dietetic supplementation
  We investigate whether an Arabinoxylan enriched crackers consumption for 4 weeks had some effects on weight loss in obese or overweight subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Muggia, Medicine, Principal Investigator — IRCCS Policlinico San Matteo Foundation
Locations (2):
- Italy (2):
  - IRCCS Policlinico San Matteo Foundation, Pavia, Pavia
  - Internal Medicine Department, Clinica Medica II, IRCCS San Matteo Foundation, Pavia, PV

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giulia Falchi A, Grecchi I, Muggia C, Palladini G, Perlini S. Effects of a Bioavailable Arabinoxylan-enriched White Bread Flour on Postprandial Glucose Response in Normoglycemic Subjects. J Diet Suppl. 2016 Nov;13(6):626-33. doi: 10.3109/19390211.2016.1156798. Epub 2016 Apr 6. PMID 27049812